CLINICAL TRIAL: NCT04248166
Title: Diagnosis of Thyroid Cancer Using Photoacoustic Imaging
Brief Title: Thyroid Cancer and Photoacoustic Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Pohang University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dong Jun Lim, Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KC15DISI0276
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Thyroid Cancer; Thyroid Nodule
Keywords: Thyroid cancer; Photoacoustic imaging
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Photoacoustic imaging — 1. Photoacoustic image of thyroid nodule is obtained by using probe of photoacoustic imaging equipment and image data and data are stored in the device.
  2. The patient's examination is the same as the general ultrasound, and the patient is asked to hold his breath for about 3-4 seconds to get the photoacoustic image.

SUMMARY:
The aim of this study was to evaluate the usefulness of photoacoustic imaging in thyroid nodules. In addition, we would like to confirm the relationship between the results of photoacoustic imaging and histopathologic findings when thyroid nodules were diagnosed as thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* All thyroid nodule identified as benign or as thyroid cancer

Exclusion Criteria:

* Patient refuses to participate in the study or withdraws consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Photoacoustic analysis of thyroid nodule and thyroid cancer | As soon as the photoacoustic test was performed
  Photoacoustic intensity of each chromophore (deoxyhemoglobin, oxyhemoglobin, lipid, water) obtained from ROI (region of interest) of photoacoustic image

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided